CLINICAL TRIAL: NCT02749604
Title: Ejaculatory Sparing vs. Non-ejaculatory Sparing GreenLightTM Laser Photoselective Vaporization of the Prostate (PVP): A Randomized Double Blind Sexual and Urodynamic Assessment
Brief Title: Ejaculatory Sparing vs. Non-ejaculatory Sparing GreenLight Laser Photoselective Vaporization of the Prostate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elshal, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mans 4-5-2016
Record Dates: First submitted 2016-04-20; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-ejaculatory sparring PVP (Active Comparator): Greenlight laser photoslective vaporization of the prostate
  Interventions: Procedure: Non-ejaculatory sparring PVP
- Ejaculatory sparring PVP (Experimental): Greenlight laser photoslective vaporization of the prostate with preservation of the ejaculatory hood
  Interventions: Procedure: Ejaculatory sparring PVP

INTERVENTIONS:
Procedure: Non-ejaculatory sparring PVP — Greenlight laser photoslective vaporization of the prostate
  Arms: Non-ejaculatory sparring PVP
Procedure: Ejaculatory sparring PVP — Greenlight laser photoslective vaporization of the prostate with preservation of the ejaculatory hood
  Arms: Ejaculatory sparring PVP

SUMMARY:
GreenLight laser PVP currently gains wide acceptance as a minimally invasive treatment for benign prostate enlargment and the emergence of ejaculatory sparing techniques made it feasible to get both benefits: relief of lower urinary tract symptoms and preservation of ejaculation. However evaluation of actual infravesical de-obstruction following such techniques remains a grey zone in the literature without an objective assessment of the degree of de-obstruction. Furthermore, the impact of maintaining ejaculation on different domains of the sexual function using comprehensive assessment tools was not compared in ejaculatory sparring vs. non-ejaculatory sparring approaches.

DETAILED DESCRIPTION:
I- Introduction:

Benign prostatic enlargement is one of the most prevalent disorders in aging men and may develop into benign prostatic obstruction (BPO) causing a significant effect on the quality of life (QoL). Clinical manifestations of BPO include a variety of lower urinary tract symptoms (LUTS) that can be classified into voiding symptoms or storage symptoms.

Laser prostatectomy includes two major technical principles; enucleation of the adenoma from the surrounding capsule or laser ablation of the adenoma. GreenLight laser (532-nm laser) and Holmium: Yttrium-Aluminum-Aarnet (Ho:YAG) laser (2100 nm) are commonly used nowadays. However, TURP remains the gold standard modality of treatment.

Ejaculation is one of the fundamental domains of male sexual functions. It is well established that ejaculation disturbances, either anejaculation or loss of antegrade ejaculation, are almost inevitable adverse effects of prostate surgery especially TURP. A problem which also associates prolonged use of α-adrenoreceptros blockers. Such adverse event can be the reason why patients may choose to avoid surgical treatment.

This ejaculatory dysfunction can be attributed, according to current theory of ejaculation, to the loss of bladder neck function after resection. However, many recent studies demonstrated that bladder neck closure may not have such important role in maintaining antegrade ejaculation. Recent techniques had been developed to preserve ejaculation including ejaculatory hood sparing technique, prostatic urethral lift and the Rezum System ( convective water vapor energy).

Ejaculatory hood was defined as paracollicular and supracollicular tissue present 1 cm proximal to the verumontanum. Hermabessiere et al. used dynamic transrectal ultrasound (TRUS) findings after TURP to demonstrate that the ejaculate is directly expelled into the infra-montanal urethra with a direct closure mechanism of the paracollicular and supracollicular tissue without previous ballooning of the prostatic urethra.

Various studies were published highlighting this ejaculation preserving technique and its impact on relieving LUTS. Alloussi et al. conducted ejaculatory preserving TURP (epTURP) on total number of 89 patients during which the ejaculatory hood area was preserved and was not affected by cutting or coagulation. Antegrade ejaculation was preserved in 90% of patients at 3 months with significant improvement of LUTS and only 12.7% of cases needed a second session for bladder neck contracture after 60 months.

GreenLight laser PVP is now challenging TURP as the standard treatment for lower LUTS caused by BPH for its many advantages e.g. short learning curve, a shorter period of postoperative bladder catheterization, lower levels of retrograde ejaculation and low indices of postoperative hematuria etc. Recently, with the introduction of the latest generation of the GreenLight laser (XPS), greenlight PVP using XPS system proved to be non inferior to TURP in reducing LUTS secondary to BPH with all the advantages of laser. [GOLIATH TRIAL].

Tabatabaei S et al. described the ejaculation preserving PVP (EP-PVP) technique applied to 160 patients and presented its outcomes. Postoperative ejaculatory function evaluation showed that 56% patients had normal antegrade ejaculation, 30.6% patients had diminished ejaculation, and 13.4% patients suffered no ejaculation. Post voiding residual urine (PVR) and peak urinary flow rate (Qmax) showed significant improvement. Overall, EP-PVP technique was successful in preserving ejaculatory function in 86.6% of patients, without compromising LUTS outcomes.

Most of published similar studies relied on degree of reduction of International prostate symptoms score (IPSS), PSA, PVR and uroflowmetry to assess the improvement of LUTS following ejaculatory preserving prostate surgery, without actual functional assessment of degree of deobstruction via urodynamic investigations.

Pereira-Correia JA et al. conducted a prospective urodynamic based trial comparing TURP and GreenLight laser PVP in total number of 20 patients over 2 years. In this study the older generation of the GreenLight laser (HPS) was utilized and conventional PVP technique was applied looking for the urodynamic changes between Greenlight PVP and TURP. They reported that high-power PVP can achieve and maintain the same results as TURP over a period of 24 months as regards improvement of infravesical obstruction evidenced by reduction of mean micturition pressure and bladder outlet obstruction index (BOOI).

GreenLight laser PVP currently gains wide acceptance and the emergence of ejaculatory sparing techniques made it feasible to get both benefits: relief of LUTS and preservation of ejaculation. However evaluation of actual infravesical deobstruction following such techniques remains a grey zone in the literature without an objective assessment of the degree of deobstruction. Furthermore, the impact of maintaining ejaculation on different domains of the sexual function using comprehensive assessment tools was not compared in ejaculatory sparring vs. non-ejaculatory sparring approaches.

II- Aim of the work

In this study, we planned to compare ejaculatory sparing and non-ejaculatory sparing (conventional) GreenLightTM Laser PVP using both subjective and objective assessment tools for the degree of deobstruction. Furthermore, the impact of both techniques on ejaculation and its secondary effect on orgasm perception and different domains of sexual function will be thoroughly assessed.

III- Patients and methods

III.1. Study design:

A randomized controlled clinical trial

Trial registration: ClinicalTrials.gov ID:

III.2. Target population:

In Prostate Unit, Mansoura urology and nephrology center, sexually active patients presented with LUTS secondary to BPO who failed medical treatment will be scheduled for GreenLightTM Laser PVP. BPH surgical candidates are patients presented with LUTS secondary to BOO due to BPH who failed medical treatment with IPSS score >15 and Peak urinary flow rate Qmax < 15 ml/min with at least 125 ml voided volume.

Legible subjects fulfilling inclusion criteria will be included in a randomized clinical trial and will be asked to sign an informed consent form according to Good Clinical Practice and the Declaration of Helsinki.

III.3. Patients' allocation:

Patients will be allocated into 2 groups. In the 1st one, patients will undergo regular non ejaculatory sparing GreenLightTM Laser PVP (Group I), while in the 2nd group (Group II); ejaculatory sparing technique will be applied. Patients are asked to sign the informed consent for participation in the study.

III.4.Methodology:

II.4.a. Intervention All laser surgeries will be performed or supervised by a single surgeon with large experience with laser prostate surgery. Procedures will be performed with the patient under general or regional anesthesia. Normal saline will be used as an irrigant. The GreenLight (532 nm) laser generator (XPS) will be used with our previously described technique for Group I. A side-to-side sweeping technique was used with the side firing fiber moving from the area of the bladder neck to approximately the level of the verumontanum. As much as possible, the end point of the laser procedure was a TURP-like cavity lined by capsular fibers, as judged by the operator.

For Group II, similar equipment will be used and steps of PVP will be similarly performed. However the procedure starts by marking of the ejaculatory hood; paracollicular and supracollicular tissue present almost 1 cm proximal to the verumontanum using the Co-Ag mode of the laser (40W). The obstructing prostate tissue will be vaporized sparing the ejaculatory hood without vaporization or coagulation at the marked hood area.

III.4.b. Assessment tools:

Ejaculatory domain of Male sexual health questionnaire (Ej-MSHQ) 16 will be used for detailed assessment of the impact of each procedure on ejaculatory function and subsequently the impact of reported ejaculatory changes on orgasm perception. This domain entails seven questions assessing ejaculatory frequency, latency, volume, force, pain, pleasure, and dry ejaculation. Each question has a score from 1 to 5 (best function) and the outcome of each question is considered significantly impaired once equals 2 or less. A total Ej-MSHQ score of good ejaculatory function was considered for a range from 28-35, average from 22 to 27 and ejaculatory dysfunction for score less than 22 .

International index of erectile function-15 (IIEF-15) 5 ; each of the five domains (EF, orgasm, desire, intercourse satisfaction and overall satisfaction) will be assessed and the degree of change from baseline to the last follow up will be depicted. EF domain is a 30 points score and normal EF is considered for score more than 25.

Urinary outcome evaluation will be done using IPSS (International prostate symptom score), QOL (quality of life), Q.max (maximum flow rate) and PVR (post void residual urine estimation).

Urodynamic evaluation will be performed in accordance with the standards recommended by the International Continence Society.

IV. Follow up:

Patients will be evaluated at baseline and will be followed post procedure at 2 weeks, one, four and twelve months interval. In the first and second visits patients will be assessed for urinary function and once their voiding parameters deemed satisfactory, they will be counseled to resume their sexual activity as before. Patients will be thoroughly evaluated at subsequent visits for both urinary and sexual outcome parameters (4 and 12 months' visits)

V.1. Randomization& masking:

The randomization process was performed using computer-generated random tables in a 1:1 ratio. Patients were randomly assigned to the study groups on the day of the surgery, once the patient signs the informed consent for participation in the study. We randomly assigned patients to one of our treatment groups by means of stratified-blocked randomization across two strata derived from predetermined size grouping (30-55ml and 55-80ml) and two strata derived from preoperative medication (alpha blockers vs. non alpha blockers user).

This method ensured parity among our two treatment groups. In each stratum, given two possible block lengths of two and four respectively, with a random number generator giving numbers uniformly distributed between 0 and 1, we selected a block length of two for random numbers lower than 0.5 or a block length of four otherwise. Variation of the block sizes prevented the surgeon from guessing what the next treatment will be; it makes it difficult (although not impossible) to break the treatment code.

V.2. Blinding:

The surgeon knew the randomly assigned laser procedure for each patient in the operating room. All patients, nurses performing urine flow studies/ addressing the questionnaires, and physician doing the urodynamic studies will be blinded to the type of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible in the study, patient must fulfill the following criteria:

  1. Age ≥ 50 years
  2. ASA (American society of anesthesiologists) score ≤3.
  3. TRUS estimated prostate weight 30-80 grams.
  4. Sexually interested and having continuous relationship with the same partner (interested).
  5. BOOI (bladder outlet obstructing index) ≥ 20 as per pressure flow study

Exclusion Criteria:

* Patients with any of the following are to be excluded:

  1. Preoperative sexual or ejaculatory disturbances or pelvic pain syndrome
  2. Documented or suspected prostate cancer (significantly elevated PSA, positive biopsy for prostate cancer guided by TRUS)
  3. Neurological disorders that can affect potency and ejaculation e.g. long standing uncontrolled DM (> 10 years) cerebral stroke, Parkinsonism
  4. Active urinary tract infection
  5. Urodynamic changes consistent with urethropathy or detrusor hypocontractility
  6. Previous pelvic surgeries
  7. History of pelvic radiotherapy

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-09 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
ejaculatory function | 4 months
  the ability to maintain ejaculatory function as depicted by Ej-MSHQ score

SECONDARY OUTCOMES:
Bladder outlet obstruction index | 4 months
  Urodynamic study looking at the dynamics of urine flow for assessment of the degree of de-obstruction
International index of erectile function-15 | 4 months
  questionnaire assessing different aspects of sexual function

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshal, Principal Investigator — Mansoura University
Locations (1):
- Urology and nephrology center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided